CLINICAL TRIAL: NCT04010331
Title: A 8 Weeks, Randomized, Double-blind, Placebo-controlled Human Trial to Evaluate the Efficacy and Safety of Nokyong Mixture Extract(CME-PI) on Promotion of Immunity
Brief Title: Efficacy and Safety of Nokyong Mixture Extract(CME-PI) on Promotion of Immunity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DC-PI-CME
Record Dates: First submitted 2019-07-03; First posted 2019-07-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Immunity
Keywords: Nokyong

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nokyong Mixture Extract(CME-PI) group (Experimental): 2 times a day, 2 capsule for 1 time, after breakfast/dinner meal(1.4g/day, Nokyong Mixture Extract(CME-PI) 1 g/day)
  Interventions: Dietary Supplement: Nokyong Mixture Extract(CME-PI)
- Placebo group (Placebo Comparator): 2 times a day, 2 capsule for 1 time, after breakfast/dinner meal(1.4g/day, Nokyong Mixture Extract(CME-PI) 0 g/day)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Nokyong Mixture Extract(CME-PI) — 2 times a day, 2 capsule for 1 time, after breakfast/dinner meal, for 8 week
  Arms: Nokyong Mixture Extract(CME-PI) group
Dietary Supplement: Placebo — Placebo for 8 week
  Arms: Placebo group

SUMMARY:
This study was conducted to investigate the efficacy and Safety of Nokyong Mixture Extract(CME-PI) on Promotion of Immunity

DETAILED DESCRIPTION:
This study was a 8 weeks, randomized, double-blind, placebo-controlled human trial. 80 subjects were randomly divided into Nokyong Mixture Extract(CME-PI) group or placebo group. The investigators measured Natural Killer cell activity, Cytokines(IL-2, IL-12, IFN-γ, TNF-α), questionnaire scores of upper airway infection.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women over 50 years
* After fully hearing and fully understanding this clinical trials, those who agree to voluntarily decide to participate and to comply with the notice

Exclusion Criteria:

* If screening shows that the white blood cell(WBC) is less than 3000/㎕ or more than 8000/㎕
* Those who received influenza vaccination within 3 months before the screening
* Those who have a body mass index(BMI) of less than 18.5 kg / m^2 or greater than 35 kg / m^2 at the screening
* Those who have a clinically significant acute or chronic cardiovascular system, endocrine system, immune system, respiratory system, liver biliary system, kidney and urinary system, neuropsychiatry, musculoskeletal system, inflammatory and hematologic
* Those who take a medication or health function food that affects your promotion of immunity within 1 month prior to the screening
* Those who have received antipsychotic medication within 3 months before screening
* Those who alcoholic or drug abuse suspected
* Those who participated in other clinical trials within 3 months before screening
* Laboratory test by show the following results

  * Aspartate Transaminase(AST), Alanine Transaminase(ALT) > Reference range 3 times upper limit
  * Serum Creatinine > 2.0 mg/dL
* Pregnancy or breast feeding
* Those who doesn't accept the implementation of appropriate contraception of a childbearing woman
* Principal Investigator judged inappropriate for participation in study because of Laboratory test result, etc.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-03-06 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-05-30 (Actual)

PRIMARY OUTCOMES:
Changes of Natural Killer cell activity | 8 weeks
  Natural Killer cell activity was measured in study baseline and 8 week. A ratio of effector cell and target cell was 50:1, 25:1, 12.5:1.
  (Experimental - Effector Spontaneous - Target Spontaneous) / (Target Maximum - Target Spontaneous) × 100

SECONDARY OUTCOMES:
Changes of Cytokines | 8 weeks
  For blood Cytokines analysis, collect 3 ml of blood in one SST tube for 5 ml, leave at room temperature for 30 minutes for clotting, after then centrifuge at 3000 rpm (or 2000 xg) for 10 minutes.
  Inspection item were IL-2, IL-6, IL-12, IFN-γ, TNF-α.
Changes of Upper respiratory infection questionnaire score | 8 weeks
  The upper respiratory infection questionnaire will investigate the occurrence of symptoms of upper respiratory infections (or symptoms), the score by symptom, the duration (days), and survey on the day of visit (1st, 2nd and 3rd visits).
  The questionnaire items were classified into three groups according to whether or not the symptoms of upper respiratory infections (or symptoms) occurrence (yes or no), the types of symptoms (sore throat, rhinorrhea, nasal obstruction, sneezing, hoarseness, myalgia, earache, fever, headache, cough, sputum, dyspnea, diarrhea, nausea, vomiting)and symptoms level (0 if no symptoms, 1 if slightly, 2 if normal, 3 severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea